CLINICAL TRIAL: NCT02808546
Title: The Risk Factors of Symptomatic Gallbladder Stone: Age-Sex Matched Case-control Study Performed in Single Institute
Status: Completed | Type: Observational
Sponsor: Cheju Halla General Hospital (Other)
Responsible Party: Principal Investigator, Byung Hyo Cha, MD, Gastroenterology Consultant, Representative of Digestive Disease Center, Cheju Halla General Hospital
Other Study IDs: 2015-L01-01
Record Dates: First submitted 2016-06-15; First posted 2016-06-21 (Estimated); Last update posted 2016-06-21 (Estimated); Status verified 2016-06

CONDITIONS: Gallstone
Keywords: Gallbladder stone; Risk factor; Case-control study; Obesity; Hypertension; Alcohol consumption
MeSH Terms: conditions — Gallstones; Cholecystolithiasis; Obesity; Hypertension; Alcohol Drinking

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Case Group: All the patients who were diagnosed as gallbladder stone disease with definite clinical symptoms and underwent cholecystectomy in Cheju Halla General Hospital, Jeju, Korea during 2009-2013
- Control Group: Control group was determined as 1:1 age-sex matched subjects selected from the participants without GBS among Health Promotion Center in the same institute and periods.

SUMMARY:
The main purpose of this study is to investigate the region-specific cause of gallbladder stone incidence in Jeju Self-Governing Province, Korea.

DETAILED DESCRIPTION:
Investigators performed the epidemiologic study to uncover the reason of relatively higher incidence of Gallbladder cancer in small isolated island, Jeju island, one of small province among 11 self governing area in South Korea. Tow studies, including descriptive epidemiology and analytic epidemiology using case-control study, some risk factors were obtained regarding Gallbladder cancer development in this area. Old age, female, and gallstone were potential risk factors and alcohol consumption was preventive factors. So authors decided to evaluate the relationship between alcohol and gallbladder stone in order to how much portion of causal relationship they have with gallbladder cancer. So this study was designed to investigate the relationship between gallbladder stone and alcohol consumption then performed clinical based case-control study with age-sex matching to each subjects.

ELIGIBILITY:
Case group

Inclusion Criteria:

* Clinical diagnosis of gallstone disease after cholecystectomy.

Exclusion Criteria:

* Ambiguous diagnosis cases for gallbladder stone.
* Incomplete medical record.

Control group

Inclusion Criteria

* Healthy examinees in Health Promotion Center in same Institute
* Eligible cases of abdominal ultrasound(US) or computed tomography(CT)

Exclusion Criteria

* The case who was diagnosed as asymptomatic gallstone on abdominal US

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Case group was enrolled from the patients who were diagnosed as gallbladder stone disease with definite clinical symptoms and underwent cholecystectomy in Cheju Halla General Hospital, Jeju, Korea during 3 years (2009-2012). And control group was determined as 1:1 age-sex matched subjects selected from the participants without GBS among Health Promotion Center in the same institute and periods.
Sampling Method: Non-Probability Sample
Enrollment: 342 (Actual)
Dates: Start 2009-01; Primary Completion 2013-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Alcohol consumption | Through study completion, an average of 1 year
  Standard Dose Drink per week was used to compare the amount of alcohol consumption of each subjects

SECONDARY OUTCOMES:
Obesity | Through study completion, an average of 1 year
  Obesity was defined as cases were scored more than 25 kg/square meter of Body Mass Index

CONTACTS AND LOCATIONS:
Overall Officials: Byung Hyo Cha, M.D., Principal Investigator — Gastroenterology Consultant

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Banim PJ, Luben RN, Bulluck H, Sharp SJ, Wareham NJ, Khaw KT, Hart AR. The aetiology of symptomatic gallstones quantification of the effects of obesity, alcohol and serum lipids on risk. Epidemiological and biomarker data from a UK prospective cohort study (EPIC-Norfolk). Eur J Gastroenterol Hepatol. 2011 Aug;23(8):733-40. doi: 10.1097/MEG.0b013e3283477cc9. PMID 21623190
- [Background] Cha BH. Epidemiological Characteristics of Gallbladder Cancer in Jeju Island: A Single-Center, Clinically Based, Age-Sex-Matched, Case-Control Study. Asian Pac J Cancer Prev. 2015;16(18):8451-4. doi: 10.7314/apjcp.2015.16.18.8451. PMID 26745100
- [Background] Chow WH, McLaughlin JK, Menck HR, Mack TM. Risk factors for extrahepatic bile duct cancers: Los Angeles County, California (USA). Cancer Causes Control. 1994 May;5(3):267-72. doi: 10.1007/BF01830247. PMID 8061176
- [Background] Little TJ, Horowitz M, Feinle-Bisset C. Role of cholecystokinin in appetite control and body weight regulation. Obes Rev. 2005 Nov;6(4):297-306. doi: 10.1111/j.1467-789X.2005.00212.x. PMID 16246215
- [Background] Randi G, Franceschi S, La Vecchia C. Gallbladder cancer worldwide: geographical distribution and risk factors. Int J Cancer. 2006 Apr 1;118(7):1591-602. doi: 10.1002/ijc.21683. PMID 16397865
- [Background] Stinton LM, Shaffer EA. Epidemiology of gallbladder disease: cholelithiasis and cancer. Gut Liver. 2012 Apr;6(2):172-87. doi: 10.5009/gnl.2012.6.2.172. Epub 2012 Apr 17. PMID 22570746